CLINICAL TRIAL: NCT05624853
Title: A Randomized, Active-controlled, Parallel, Open-label, Multicenter, Phase 4 Study to Compare the Efficacy and Safety of Pregabalin Sustained Release Tablet and Pregabalin Immediate Release Capsule in Type II Diabetic Patients With Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC042
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Neuropathic Pain; Diabetes Mellitus, Type 2
Keywords: pregabalin sustained release tablet
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus, Type 2 | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregabalin sustained release tablet (Experimental): pregabalin sustained release tablet 150mg qd for 8weeks
  Interventions: Drug: pregabalin sustained release tablet
- pregabalin immediate release capsule (Active Comparator): pregabalin immediate release capsule 75mg bid for 8weeks
  Interventions: Drug: pregabalin immediate release capsule

INTERVENTIONS:
Drug: pregabalin sustained release tablet — pregabalin sustained release tablet 150mg qd for 8weeks
  Arms: pregabalin sustained release tablet
Drug: pregabalin immediate release capsule — pregabalin immediate release capsule 75mg bid for 8weeks
  Arms: pregabalin immediate release capsule

SUMMARY:
This study is to compare the efficacy and safety of pregabalin sustained release tablet and pregabalin immediate release capsule in type II diabetic patients with peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 19 years, < 75 years
2. VAS score for diabetic peripheral neuropathy pain ≥ 30
3. Patients who have been administering pregabalin immediate release capsule 150 mg/day for more than 4 weeks
4. Type II DM patient and HbA1c ≤ 10 %
5. Written informed consent

Exclusion Criteria:

1. Patient with hypersensitivity to pregabalin
2. Patient on anti-epileptic drugs
3. Patients with pain caused by other factors than diabetic peripheral neuropathy
4. Patients undergoing eGFR <30 mL/min/1.73 m2 (MDRD) at screening
5. AST(Aspartate Aminotransferase) or ALT(Alanine Aminotransferase) level ≥ 3x ULN (upper limit of normal range) or active liver disease
6. Drug-abusing patient
7. Severe depression or uncontrolled abnormal mood and behavioral changes
8. Pregnant and breast-feeding woman
9. Patients who participated in other clinical trials for investigational products within 30 days of screening
10. Patients deemed to be ineligible to participate in the trial by investigator

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 in Visual Analogue Scale(VAS) | Baseline/Week 8

SECONDARY OUTCOMES:
Change from baseline to week 8 in Quality of Life(EQ-5D) | Baseline/Week 8
Change from baseline to week 8 in Patients Global Impression of Change(PGIC) | Baseline/Week 8
Change from baseline to week 8 in Clinician Global Impression of Change(CGIC) | Baseline/Week 8
Change from baseline to week 8 in Daily Sleep Interference Scale(DSIS) | Baseline/Week 8
Change from baseline to week 8 in Morisky Medication Adherence Scale 8-item version(MMAS-8) | Baseline/Week 8
Dose and frequency of Rescue medication(Acetaminophen) | Baseline/Week 8
Number and proportion of subjects with adverse event | Baseline/Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bon Jeong Ku, Principal Investigator — Chungnam National University Hospital
Locations (8):
- South Korea (8):
  - Dankook University Hospital, Cheonan, Chungcheongnam-do
  - Catholic University of Korea's Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Chungnam National University Sejong Hospital, Sejong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joung KH, Kim TN, Ku EJ, Lee SS, Yoo WS, Park KS, Kwon SK, Ku BJ. A phase 4 randomized active-controlled clinical study to compare the efficacy and safety of sustained-release pregabalin with immediate-release pregabalin in type 2 diabetic patients with peripheral neuropathic pain. J Diabetes Complications. 2024 Aug;38(8):108809. doi: 10.1016/j.jdiacomp.2024.108809. Epub 2024 Jul 14. PMID 39018898